CLINICAL TRIAL: NCT02756039
Title: Tagrisso Tablets Clinical Experience Investigation (All Case Investigation)
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5160C00025
Record Dates: First submitted 2016-04-28; First posted 2016-04-29 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: All Patients Treated With the Product

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Clinical experience investigation (CEI) is to be conducted to confirm the following to characterise safety and efficacy of Tagrisso Tablets in actual clinical use.

1. Incidence of adverse drug reactions (ADRs) in actual clinical use
2. Factors which may affect safety and efficacy of the product (especially analysis of the incidence and risk factors of interstitial lung disease (ILD) events)
3. Information of ADRs not expected from "Precautions for Use" of the package insert in Japan

ELIGIBILITY:
Inclusion Criteria:

* patients treated with the product

Exclusion Criteria:

* No Account (NA)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients treated with the product will be enrolled in the investigation.
Sampling Method: Probability Sample
Enrollment: 3494 (Actual)
Dates: Start 2016-05-25 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions (ADRs) in actual clinical use | Up to 12 months
  Presence/absence of adverse events (AEs) [any undesirable or unintentional signs (including laboratory abnormalities), symptoms, or diseases whether or not considered causally related to the product] reported during the observation period However, deterioration of a pre-existing lung cancer lesion and lung cancer death should not be reported as an AE.

CONTACTS AND LOCATIONS:
Locations (47):
- Japan (47):
  - Research Site, Aichi
  - Research Site, Akita
  - Research Site, Aomori
  - Research Site, Chiba
  - Research Site, Ehime
  - Research Site, Fukui
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Gifu
  - Research Site, Gunma
  - Research Site, Hiroshima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Ishikawa
  - Research Site, Kagawa
  - Research Site, Kagoshima
  - Research Site, Kanagawa
  - Research Site, Kochi
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Mie
  - Research Site, Miyagi
  - Research Site, Miyazaki
  - Research Site, Nagano
  - Research Site, Nagasaki
  - Research Site, Nara
  - Research Site, Niigata
  - Research Site, Numakunai
  - Research Site, Okayama
  - Research Site, Okinawa
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Saga
  - Research Site, Saitama
  - Research Site, Shiga
  - Research Site, Shimane
  - Research Site, Shizuoka
  - Research Site, Tochigi
  - Research Site, Tokushima
  - Research Site, Tokyo
  - Research Site, Tottori
  - Research Site, Toyama
  - Research Site, Wakayama
  - Research Site, Yamagata
  - Research Site, Yamaguchi
  - Research Site, Yamanashi

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5160C00025&attachmentIdentifier=a861804d-5228-447d-b85c-41680e2c43ba&fileName=AZ_Synopsis_TAG_E_final.pdf&versionIdentifier=